CLINICAL TRIAL: NCT03364257
Title: National, Single-arm Clinical Study on iDTECT™ Blood Performance to Identify Viral or Bacterial Pathogens in Febrile Neutropenic Patients With Suspected Infection
Brief Title: iDTECT Blood Performance for the Identification of Viral or Bacterial Pathogens in Febrile Neutropenic Patients
Acronym: IDENTIFY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pathoquest (Industry)
Responsible Party: Sponsor
Other Study IDs: PTQ-02
Record Dates: First submitted 2017-11-28; First posted 2017-12-06 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Febrile Neutropenia; Acute Leukemia; Stem Cell Transplantation; Infection
Keywords: metagenomic; infection; diagnosis
MeSH Terms: conditions — Febrile Neutropenia; Infections; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: iDTECT Blood — Next generation sequencing-based shot-gun metagenomic test for the diagnosis of viral or bacterial infections using blood samples

SUMMARY:
Prospective, multicentre French observational study assessing the performance and medico-economic utility of iDTECT Blood versus conventional microbiologic diagnosis in patients with febrile neutropenia

DETAILED DESCRIPTION:
Febrile neutropenic patients suspected of sepsis will follow the conventional infectious diagnosis work-up over the entire observation period, and will be tested in addition with iDTECT Blood on Study Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 5 years and weight > 16 Kg
2. Patients having signed the written study informed consent form (ICF) prior to any study-mandated procedure. For children/adolescents: ICF obtained from both children's parents/ legal representative prior to any study-mandated procedure, and in addition for adolescents (13-17 years): assent form to be signed
3. Patient presenting severe neutropenia (absolute neutrophil count < 0.5 Giga/L) anticipated to be long lasting (> 10 days) following intensive chemotherapy for acute myeloid or lymphoid leukaemia (AML or ALL) or myelodysplastic syndrome or in the context of hematopoietic stem cells transplantation
4. Febrile episode (oral temperature > 38.3°C once, or 2 measures > 38.0°C taken 2h apart).

Exclusion Criteria:

1. Known HIV infection or AIDS diagnosis
2. Already microbiologically confirmed infection
3. Patient status preventing the study test to be performed
4. Patient with an obvious infectious disease diagnosis requiring minimal additional microbiological documentation or confirmation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with chemotherapy for Acute Leukaemia (AL) or Myelodysplastic Syndrome (MDS) or in the context of hematopoietic stem cell transplantation (HSCT), presenting a febrile neutropenic episode and suspected of infection
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of detection of clinically relevant bacterial or viral pathogen (CRBV) by iDTECT™ Blood as compared to conventional microbiological methods at inclusion | 7 months
  Sensitivity, specificity, negative predictive value, positive predictive value at inclusion

SECONDARY OUTCOMES:
Antiobiotic use | 9 months
  Type of antibiotic, duration of antibiotic course

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hospital Necker, Paris
  - Hospital Robert Debré, Paris
  - Hospital Salpétrière, Paris
  - Hospital Trousseau, Paris
  - Hosptial Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: Undecided